CLINICAL TRIAL: NCT01174394
Title: A Randomized, Assessor-blind, Controlled Trial of Electroacupuncture Combined With Antidepressants in Treating Patients With Post-stroke Depression
Brief Title: Electroacupuncture Combined With Antidepressants for Post-stroke Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Tung Wah Hospital (Other); Kowloon Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Zhang Zhang-Jin, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW 10-211
Record Dates: First submitted 2010-07-29; First posted 2010-08-03 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Depression; Stroke
Keywords: Acupuncture; Post Stroke Depression; Depressive Disorder; Cardiovascular Accident; Stroke; Apoplexy; CVA
MeSH Terms: conditions — Depression; Stroke; Depressive Disorder | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DCEAS (Experimental): Body electroacupuncture plus dense cranial electroacupuncture stimulation (DCEAS)
  For those who were currently under antidepressant treatment, they would continue the existing treatment regimens. For those who were not medicated at the time of trial, fluoxetine (FLX) was given at an initiate dose of 10 mg/day and escalated to an optimal dose within one week, based on individual response, but the maximum dose was set at 40 mg/day.
  Interventions: Procedure: DCEAS (Hwato®/ Dongbang®); Procedure: Body electro-acupuncture (Hwato®/ Dongbang®); Drug: Fluoxetine
- n-CEA (Placebo Comparator): Body electroacupuncture plus non-invasive cranial electroacupuncture (n-CEA)
  For those who were currently under antidepressant treatment, they would continue the existing treatment regimens. For those who were not medicated at the time of trial, fluoxetine (FLX) was given at an initiate dose of 10 mg/day and escalated to an optimal dose within one week, based on individual response, but the maximum dose was set at 40 mg/day.
  Interventions: Procedure: Body electro-acupuncture (Hwato®/ Dongbang®); Procedure: n-CEA (Strietberger®); Drug: Fluoxetine

INTERVENTIONS:
Procedure: DCEAS (Hwato®/ Dongbang®) — Upon insertion of acupuncture needles, dense cranial electro-acupuncture stimulation (DCEAS), is directly delivered on a density of cranial acupoints (in general 6-8 pairs) located on the frontal, parietal, and temporal scalp areas.
  Other Names: Hwato®; Dongbang®
  Arms: DCEAS
Procedure: Body electro-acupuncture (Hwato®/ Dongbang®) — Both study arms received body electroacupuncture on both sides of ipsilateral limb pairs: Hegu (LI4) and Quchi (LI11) , Zusanli (ST36) and Taichong (LR3). Electrical stimulation as DCEAS is applied.
  Other Names: Hwato®; Dongbang®
Procedure: n-CEA (Strietberger®) — Streitberger's non-invasive acupuncture needles were applied to serve as sham control at the same cranial acupoints and the same stimulation modality, except that the needles only adhere to the skin instead of insertion
  Other Names: Strietberger®
  Arms: n-CEA
Drug: Fluoxetine — Subjects of both study arms received orally administered SSRIs for 4 weeks in an open manner. For those who were currently under antidepressant treatment, they would continue the existing treatment regimens. For those who were not medicated at the time of trial, fluoxetine (FLX) was given at an initiate dose of 10 mg/day and escalated to an optimal dose within one week, based on individual response, but the maximum dose was set at 40 mg/day.
  Other Names: Prozac; Sarafem; Fontex; Zactin; Lovan; Fluohexal; Auscap; Depreks; Floxet; Flunil; Fluox; Fluzac; Fluxen

SUMMARY:
This is a randomized, assessor-blind, placebo controlled study in post stroke depression patients. Subjects receiving antidepressant drug would be assigned to either active or placebo scalp electro-acupuncture treatment, on the hypothesis that acupuncture intervention combined with antidepressants could produce greater therapeutic effects than antidepressants alone.

DETAILED DESCRIPTION:
Mood depression is a common and serious consequence of stroke. A large proportion of stroke patients develop post-stroke depression (PSD), either in the early or late stages after stroke. Although antidepressant agents, represented by selective serotonin reuptake inhibitors (SSRIs), are recommended as first-line drugs in pharmaco-therapy of PSD, its effectiveness is limited and the clinical use is largely hampered due to broad side effects, especially on cardiovascular system. In addition, since stroke patients are often medicated with various classes of drugs, the addition of antidepressant agents may increase risk of drug-drug interactions, resulting in unexpected and unpredictable adverse events.

The objective of this proposed study is to determine whether electro-acupuncture (EA) combined with antidepressants could produce significantly greater improvement on depressive symptoms in patients with PSD compared to antidepressants alone.

In this 4-week, assessor-blind, randomized, controlled study of electro-acupuncture (EA) as additional treatment with the antidepressant drug called fluoxetine (FLX), a total of 60 patients with post-stroke depression (PSD) will be recruited. The patients will be randomly assigned to FLX (10-30 mg/day) combined with active cranial and body acupuncture (n =30) or FLX with placebo cranial and active body acupuncture (n =30) (12 sessions, 3 sessions a week). Changes in the severity of depressive symptoms over time are measured using depressive scale instruments. Clinical response and remission rates are also calculated. The study will be conducted at HKU School of Chinese Medicine, Tung Wah Hospital, and Kowloon Hospital, Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* most recently experience an ischemic or hemorrhagic stroke, documented by cerebral computed topographic scanning or magnetic resonance imaging
* develop significant depression, with a HAMD-17 score of 16 or greater

Exclusion Criteria:

* presence of severe aphasia, especially fluent aphasia
* presence of severe cognitive dysfunction, indicated the Mini-mental State Examination (MMSE) score of < 18
* had a history of psychiatric illness other than depression
* presence of another chronic disorder, including severe Parkinson's disease, cardiac disease, cancers, epilepsy, or chronic alcoholism
* impaired hepatic or renal function
* have bleeding tendency

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
HAMD-17, GDS , BI and CGI | 28-day (course of treatment)
  Depression symptoms are primarily measured using the 17-item Hamilton Depression Scale (HAMD-17) and Geriatric Depression Scale (GDS); physical outcomes will be measured using Barthel Index (BI); Clinical Global Impression (CGI) would also be measured by clinician. The measurements are carried out at the baseline, first, second and fourth week of treatment course.

SECONDARY OUTCOMES:
Clinical response, latency and adverse events | 28-day (course of treatment)
  The secondary efficacy measures include clinical response, defined as greater than or equal to 50% reduction at endpoint from baseline on HAMD-17; remission, defined as 7 points or less on HAMD-17 score; and the latency of the clinical response. The measurements are carried out at the baseline, first, second and fourth week of treatment course.
  Adverse events are assessed using the Treatment Emergent Symptom Scale (TESS) when applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang-Jin Zhang, MMed, PhD, Principal Investigator — The University of Hong Kong
Locations (3):
- Hong Kong (3):
  - Tung Wah Hospital - Rehabilitation Unit, Department of Medicine, Hong Kong
  - Kowloon Hospital - Department of Psychiatry, Kowloon
  - Kowloon Hospital - Department of Rehabilitation, Kowloon

REFERENCES:
- [Derived] Man SC, Hung BH, Ng RM, Yu XC, Cheung H, Fung MP, Li LS, Leung KP, Leung KP, Tsang KW, Ziea E, Wong VT, Zhang ZJ. A pilot controlled trial of a combination of dense cranial electroacupuncture stimulation and body acupuncture for post-stroke depression. BMC Complement Altern Med. 2014 Jul 19;14:255. doi: 10.1186/1472-6882-14-255. PMID 25038733